CLINICAL TRIAL: NCT01464099
Title: A Single Center, Randomized, Double-blind, Balanced Two-period Cross-over Trial to Test for Bioequivalence Between a Marketed NovoLog® Formulation Containing 100 U/mL Versus a New NovoLog® Formulation Containing 200 U/mL in a Combined Regimen of a Continuous Subcutaneous Infusion and a Meal-time Bolus in Subjects With Type 1 Diabetes
Brief Title: Bioequivalence of Two NovoLog® Formulations in Subjects With Type 1 Diabetes
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Novo Nordisk A/S (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: ANA-3501
Record Dates: First submitted 2011-10-31; First posted 2011-11-03 (Estimated); Last update posted 2016-10-28 (Estimated); Status verified 2016-10

CONDITIONS: Diabetes; Diabetes Mellitus, Type 1
MeSH Terms: conditions — Diabetes Mellitus; Diabetes Mellitus, Type 1 | interventions — Insulin Aspart

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Insulin aspart 100U/mL (Active Comparator)
  Interventions: Drug: insulin aspart
- Insulin aspart 200U/mL (Experimental)
  Interventions: Drug: insulin aspart

INTERVENTIONS:
Drug: insulin aspart — An initial priming dose of insulin aspart is administered, then a continuous subcutaneous insulin aspart infusion followed by a bolus of insulin aspart on top of the continuous insulin aspart infusion
  Arms: Insulin aspart 100U/mL
Drug: insulin aspart — An initial priming dose of insulin aspart is administered, then a continuous subcutaneous insulin aspart infusion followed by a bolus of insulin aspart on top of the continuous insulin aspart infusion
  Arms: Insulin aspart 200U/mL

SUMMARY:
This trial is conducted in the United States of America (USA). The aim of this trial is to evaluate the clinical performance of two formulations of insulin aspart (NovoLog®) in subjects with type 1 diabetes.

ELIGIBILITY:
Inclusion Criteria:

* Subjects with type 1 diabetes treated with insulin for at least 12 months
* BMI (Body Mass Index) between 18.0-29.0 kg/m^2
* Negative fasting C-peptide (below or equal to 0.6 ng/mL)
* HbA1c (glycosylated haemoglobin A1c) below or equal to 10.0%
* Current treatment with insulin below or equal to 1.2 U/kg/day
* Subject should be in good health based on medical history, physical examination and routine laboratory data

Exclusion Criteria:

* Any known/suspected allergies to trial medication or similar products/devices
* A subject who has proliferative retinopathy or maculopathy, and/or severe neuropathy, in particular autonomic neuropathy, as judged by the Investigator
* Clinically significant active disease of any kind
* Recurrent major hypoglycemia or hypoglycemic unawareness, as judged by the Investigator
* Blood donation (more than 500 mL) within the previous 9 weeks

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2008-06; Primary Completion 2008-11 (Actual); Study Completion 2008-11 (Actual)

PRIMARY OUTCOMES:
Area under the insulin aspart bolus concentration-time curve | From 0 and up to 12 hours post bolus dose administration
Maximum plasma concentration (Cmax) of insulin aspart | From 0 and up to 12 hours post bolus dose administration

SECONDARY OUTCOMES:
Time to maximum concentration (Tmax) of insulin aspart | From 0-12 hours post bolus dose administration
AUC (area under the curve) of insulin aspart | From -4 to 0 hours after dose administration

CONTACTS AND LOCATIONS:
Overall Officials: Global Clinical Registry (GCR, 1452), Study Director — Novo Nordisk A/S
Locations (1):
- Novo Nordisk Investigational Site, Chula Vista, California, United States

REFERENCES:
- See also: Clinical Trials at Novo Nordisk — http://novonordisk-trials.com